CLINICAL TRIAL: NCT02784067
Title: A Multicenter, Double-Blind, Placebo-Controlled Trial to Evaluate the Frequency of Genetic Sucrase-Isomaltase Deficiency Genotypes, and the Efficacy and Safety of Sucraid® (Sacrosidase) Oral Solution in Subjects With Chronic Diarrhea and Sucrase Deficiency
Brief Title: A Trial to Evaluate the Frequency of Genetic Sucrase-Isomaltase Deficiency Genotypes, and the Efficacy and Safety of Sucraid® (Sacrosidase) Oral Solution in Subjects With Chronic Diarrhea and Sucrase Deficiency
Acronym: GSID-E
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Clinical Trial Material
Sponsor: QOL Medical, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: S09A
Record Dates: First submitted 2016-05-18; First posted 2016-05-26 (Estimated); Last update posted 2017-09-25 (Actual); Status verified 2017-09

CONDITIONS: Genetic Sucrase-Isomaltase Deficiency
MeSH Terms: interventions — beta-Fructofuranosidase

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment (Experimental): Subjects randomized to the active treatment arm will take Sucraid, 2 mL (17,000 IU) with every meal or snack, administered orally following dilution with 2 to 4 ounces (60 to 120 mL) of water or milk (either cold or at room temperature). The study treatment period is one week.
  Interventions: Drug: Sucraid
- Placebo (Placebo Comparator): Subjects randomized to the placebo treatment arm will take Sucraid placebo, 2 mL (17,000 IU) with every meal or snack, administered orally following dilution with 2 to 4 ounces (60 to 120 mL) of water or milk (either cold or at room temperature). The study treatment period is one week.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sucraid — Study drug
  Other Names: Sacrosidase
  Arms: Treatment
Drug: Placebo — Sucraid placebo
  Arms: Placebo

SUMMARY:
S09A is a Phase 4, multicenter, randomized, double-blind, placebo-controlled, parallel study examining the efficacy and safety of a Sucraid (sacrosidase) Oral Solution in comparison to a placebo in 150-200 subjects with chronic diarrhea possibly attributable to sucrase deficiency.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is 16 years of age or older.
2. Subject is male or female. Women of childbearing potential must be willing to use one of the following contraception methods (for at least 10 days prior to start of study drug and for 10 to 14 days after last dose of study drug): Oral contraceptive, Injectable progestogen, Implants of levonorgestrel, Estrogenic vaginal ring, Percutaneous contraceptive patches, Intrauterine device, Sterile male partner, Double-barrier method of contraception Women of non-child bearing potential include females regardless of age with functioning ovaries and who have a current tubal ligation (Hatcher, 2004), bilateral oophorectomy, or total hysterectomy, or post-menopausal females. Note: Post-menopausal is defined as 1 year without menses with an appropriate clinical profile (e.g., age appropriate, >45 years, in the absence of hormone replacement therapy).
3. Subject has a minimum of 3 months of self-reported diarrhea (BSFS scores ≥ 5 on at least 3 days per week and ≥1 stool per day)
4. Subject has a value in the SHMBT of at least 20 ppm for hydrogen, or 12 ppm for methane or 15 ppm above a previous breath sample for the combination of both gases.
5. Subject reports that he/she experienced soft stools or diarrhea within the last 24 hours when contacted by the site 24 hours after completing the SHMBT.
6. Subject is able to read, speak, and verbally understand the English language.
7. Subject is located in the United States.
8. Subject has access to the Internet on a daily basis.
9. Subject has access to an acceptable Apple iPhone/iPad/iTouch or Android smartphone/tablet. The sponsor may choose to provide a smartphone in unusual cases (please contact sponsor to request loaner device when applicable)

Exclusion Criteria:

1. Subject has recent history of functional or chronic constipation.
2. Subject has known history of ulcerative colitis, Crohn's disease, or Celiac disease.
3. Subject has known hypersensitivity to papain, glycerol, or yeast.
4. Subject has received bovine serum in the last year.
5. Subject has previous history of Sucraid use.
6. Subject has taken any prebiotic or probiotic within 5 days prior to Visit 2 and does not agree to refrain from taking them during the study.
7. Subject is female and is pregnant, breastfeeding, or planning to become pregnant during the study.
8. Subject has known uncontrolled systemic disease.
9. Subject has prior diagnosis of Type 1 or Type 2 diabetes.
10. Subject has history of bowel resection.
11. Subject is undergoing chemotherapy for the treatment of cancer.
12. Subject has major physical or psychiatric illness within the last 6 months that in the opinion of the investigator would affect the subject's ability to complete the trial.
13. Subject has used an investigational device or investigational drug within 30 days prior to Visit 1.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-05; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Response to Sucraid and placebo in a parallel group study based on improvement in daily stool consistency, as assessed by the BSFS using SHMBT | Up to 2 years
  Response to Sucraid and placebo based on improvement in daily stool consistency, as assessed by the Bristol Stool Form Scale (BSFS) over a 1-week treatment period in subjects with chronic diarrhea and sucrase deficiency using a sucrose hydrogen methane breath test (SHMBT).

SECONDARY OUTCOMES:
Effects of Sucraid and placebo on daily assessments of Bristol Stool Form Scale | Up to 2 years
Effects of Sucraid and placebo on daily stool frequency | Up to 2 years
Effects of Sucraid and placebo on daily abdominal pain | Up to 2 years
Effects of Sucraid and placebo on daily bloating severity | Up to 2 years
The relationship between the severity of sucrase deficiency, quantified by a SHMBT | Up to 2 years
The mean improvement in the BSFS for each treatment group. | Up to 2 years
Overall frequency of the 4 most common sucrase-isomaltase deficiency genetic variants | Up to 2 years
  Overall frequency of the 4 most common sucrase-isomaltase deficiency genetic variants in comparison to the frequency in public proxy databases of broad populations.
The number of less common sucrase-isomaltase polymorphisms in this study population. | Up to 2 years
The allele frequency of the most common sucrase-isomaltase genetic variants in subjects with chronic diarrhea attributable to sucrase deficiency compared to the allele frequency in other databases | Up to 2 years
  Assess the allele frequency of the 38 most common sucrase-isomaltase genetic variants in subjects with chronic diarrhea attributable to sucrase deficiency compared to the allele frequency of sucrase-isomaltase genetic variants in the Exome Variant Server, the ExAC server, and other public proxy and private genetic databases.

REFERENCES:
- [Background] Arthur AB. Intestinal disaccharidase deficiency in children with coeliac disease. Arch Dis Child. 1966 Oct;41(219):519-24. doi: 10.1136/adc.41.219.519. No abstract available. PMID 5957725
- [Background] Bayless TM, Christopher NL. Disaccharidase deficiency. Am J Clin Nutr. 1969 Feb;22(2):181-90. doi: 10.1093/ajcn/22.2.181. PMID 4885929
- [Background] Chumpitazi BP, Robayo-Torres CC, Tsai CM, Opekun AR, Baker SS, Nichols BL, Gilger MA, Su1110 Yield of prospective disaccharidase testing in children with recurrent abdominal pain. Gastroenterology. May 2013;144(5):S-401-S402.
- [Background] Cross HS, Quaroni A. Inhibition of sucrose-isomaltase expression by EGF in the human colon adenocarcinoma cells Caco-2. Am J Physiol. 1991 Dec;261(6 Pt 1):C1173-83. doi: 10.1152/ajpcell.1991.261.6.C1173. PMID 1767818
- [Background] Czernichow B, Simon-Assmann P, Kedinger M, Arnold C, Parache M, Marescaux J, Zweibaum A, Haffen K. Sucrase-isomaltase expression and enterocytic ultrastructure of human colorectal tumors. Int J Cancer. 1989 Aug 15;44(2):238-44. doi: 10.1002/ijc.2910440209. PMID 2759730
- [Background] DeMets DL, Lan KK. Interim analysis: the alpha spending function approach. Stat Med. 1994 Jul 15-30;13(13-14):1341-52; discussion 1353-6. doi: 10.1002/sim.4780131308. PMID 7973215
- [Background] El-Chammas K, Williams S, Miranda A. Su1254 Lactase and sucrase deficiencies in pediatric subjects with chronic abdominal pain. Gastroenterology. May 2014;146(5):S-415-S416.
- [Background] Gupta SK, Chong SK, Fitzgerald JF. Disaccharidase activities in children: normal values and comparison based on symptoms and histologic changes. J Pediatr Gastroenterol Nutr. 1999 Mar;28(3):246-51. doi: 10.1097/00005176-199903000-00007. PMID 10067723
- [Background] Hatcher RA, Trussell J, Stewart F, Nelson AL, Cates W, Guest F, Kowal DD, editors. Contraceptive Technology. New York: Ardent Media, 2004:226.
- [Background] Heitlinger LA, Rossi TM, Lee PC, Lebenthal E. Human intestinal disaccharidase activities: correlations with age, biopsy technique, and degree of villus atrophy. J Pediatr Gastroenterol Nutr. 1991 Feb;12(2):204-8. PMID 1904933
- [Background] Hyams JS, Batrus CL, Grand RJ, Sallan SE. Cancer chemotherapy-induced lactose malabsorption in children. Cancer. 1982 Feb 15;49(4):646-50. doi: 10.1002/1097-0142(19820215)49:43.0.co;2-m. PMID 7055778
- [Background] Kerry KR, & Townley, R. R. Genetic aspects of intestinal sucrase-isomaltase deficiency. Australian Paediatric Journal. 1965;1:223.
- [Background] Lehmacher W, Wassmer G. Adaptive sample size calculations in group sequential trials. Biometrics. 1999 Dec;55(4):1286-90. doi: 10.1111/j.0006-341x.1999.01286.x. PMID 11315085
- [Background] Mones RL, Yankah A, Duelfer D, Bustami R, Mercer G. Disaccharidase deficiency in pediatric patients with celiac disease and intact villi. Scand J Gastroenterol. 2011 Dec;46(12):1429-34. doi: 10.3109/00365521.2011.619276. Epub 2011 Sep 22. PMID 21936724
- [Background] Murray IA, Smith JA, Coupland K, Ansell ID, Long RG. Intestinal disaccharidase deficiency without villous atrophy may represent early celiac disease. Scand J Gastroenterol. 2001 Feb;36(2):163-8. doi: 10.1080/003655201750065915. PMID 11252408
- [Background] Nichols BL Jr, Adams B, Roach CM, Ma CX, Baker SS. Frequency of sucrase deficiency in mucosal biopsies. J Pediatr Gastroenterol Nutr. 2012 Nov;55 Suppl 2:S28-30. doi: 10.1097/01.mpg.0000421405.42386.64. No abstract available. PMID 23103647
- [Background] O'Brien PC, Fleming TR. A multiple testing procedure for clinical trials. Biometrics. 1979 Sep;35(3):549-56. PMID 497341
- [Background] Osterlund P, Ruotsalainen T, Peuhkuri K, Korpela R, Ollus A, Ikonen M, Joensuu H, Elomaa I. Lactose intolerance associated with adjuvant 5-fluorouracil-based chemotherapy for colorectal cancer. Clin Gastroenterol Hepatol. 2004 Aug;2(8):696-703. doi: 10.1016/s1542-3565(04)00293-9. PMID 15290663
- [Background] Quezada-Calvillo R, Sim L, Ao Z, Hamaker BR, Quaroni A, Brayer GD, Sterchi EE, Robayo-Torres CC, Rose DR, Nichols BL. Luminal starch substrate "brake" on maltase-glucoamylase activity is located within the glucoamylase subunit. J Nutr. 2008 Apr;138(4):685-92. doi: 10.1093/jn/138.4.685. PMID 18356321
- [Background] Reed, JF. (2006) AB/BA Crossover Trials - Binary Outcome. J Modern Applied Stat Methods 5 (2): 452-457.
- [Background] Treem WR. Clinical aspects and treatment of congenital sucrase-isomaltase deficiency. J Pediatr Gastroenterol Nutr. 2012 Nov;55 Suppl 2:S7-13. doi: 10.1097/01.mpg.0000421401.57633.90. No abstract available. PMID 23103658
- [Background] Treem WR, McAdams L, Stanford L, Kastoff G, Justinich C, Hyams J. Sacrosidase therapy for congenital sucrase-isomaltase deficiency. J Pediatr Gastroenterol Nutr. 1999 Feb;28(2):137-42. doi: 10.1097/00005176-199902000-00008. PMID 9932843
- [Background] Treem WR. Congenital sucrase-isomaltase deficiency. J Pediatr Gastroenterol Nutr. 1995 Jul;21(1):1-14. doi: 10.1097/00005176-199507000-00001. No abstract available. PMID 8576798
- [Background] Treem WR, Ahsan N, Sullivan B, Rossi T, Holmes R, Fitzgerald J, Proujansky R, Hyams J. Evaluation of liquid yeast-derived sucrase enzyme replacement in patients with sucrase-isomaltase deficiency. Gastroenterology. 1993 Oct;105(4):1061-8. doi: 10.1016/0016-5085(93)90950-h. PMID 8405850
- [Background] Uhrich S, Wu Z, Huang JY, Scott CR. Four mutations in the SI gene are responsible for the majority of clinical symptoms of CSID. J Pediatr Gastroenterol Nutr. 2012 Nov;55 Suppl 2:S34-5. doi: 10.1097/01.mpg.0000421408.65257.b5. No abstract available. PMID 23103650
- [Background] Wiecek S, Wos H, Radziewicz Winnicki I, Komraus M, Grzybowska Chlebowczyk U. Disaccharidase activity in children with inflammatory bowel disease. Turk J Gastroenterol. 2014 Apr;25(2):185-91. doi: 10.5152/tjg.2014.3994. PMID 25003680